CLINICAL TRIAL: NCT05937555
Title: Professional Bladder Cancers and the Profession of Painter: Retrospective Study of the RNV3P Database Files
Brief Title: Professional Bladder Cancers and the Profession of Painter
Acronym: NEVPP
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC19.0259 - NEVPP
Record Dates: First submitted 2022-04-04; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Bladder Cancer
Keywords: painter; occupational cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

SUMMARY:
This is a retrospective study on bladder cancer in French painters' population. The French agency ANSES collected data from all occupational and environmental diseases center in a specific database called RNV3P. We selected cases of bladder cancer in painters in four centers from 01/01/2010 to 31/12/2019. Those cases were analyzed in terms of occupational exposure, histology and sociodemographics data. Comparison between different histologic types of cancer, workplaces and occupational diseases process will be done.

ELIGIBILITY:
Inclusion Criteria:

* painters
* age> 18 years
* data from one of the French occupational diseases centers
* approval letter

Exclusion Criteria:

* non-approval letter
* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: workers with occupational work tasks of painting with medical consultation for bladder cancer in a French occupational diseases center
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
histological type of bladder cancer | Inclusion ( Day 0)
  international classification of bladder cancer TNM and histology

SECONDARY OUTCOMES:
Occupational exposures | Inclusion (Day 0)
  chemical exposures and workplaces during occupational painting activities

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHRU de Brest, Brest
  - CHU de Caen, Caen
  - Ch Cherbourg, Cherbourg
  - CH le Havre, Le Havre
  - CHU de Lille, Lille
  - CHU de Rouen, Rouen